CLINICAL TRIAL: NCT04562493
Title: Comparative Effect of Transforaminal Injection of Magnesium Sulphate Versus Ozone Therapy on Oxidative Stress Biomarkers in Lumbar Disc Related Radicular Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Wael Fathy Hassan, Lecturer of Anaesthesia and pain, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMBSUREC/01122019/Hussein
Record Dates: First submitted 2020-09-03; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Effect of Drug

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magnesium sulphate group (Active Comparator): Effect of transforaminal Magnesium sulphate on oxidative stress markers and radicular pain
  Interventions: Procedure: Transforaminal Epidural injection
- Ozone Group (Experimental): Effect of transforaminal Ozone on oxidative stress markers and radicular pain
  Interventions: Procedure: Transforaminal Epidural injection
- Steroid group (Other): Effect of transforaminal steroids on oxidative stress markers and radicular pain
  Interventions: Procedure: Transforaminal Epidural injection

INTERVENTIONS:
Procedure: Transforaminal Epidural injection — Transforaminal injection will be performed under fluoroscopy guidance. The patient will be placed in the prone position and draped in the sterile manner. A 22-gauge, 3.5-inch spinal needle will be used. The selected patients will receive transforaminal epidural injection of the drug

SUMMARY:
Chronic lumbar radicular (CLR) pain is a term used to describe neuropathic pain symptoms in the distribution of a particular lumbar nerve root due to disc protrusion, spinal stenosis, facet hypertrophy, or fibrosis after previous surgery. The pathophysiology of CLR pain involves mechanical, inflammatory, and immunologic factors that affect the function of the dorsal root ganglion (DRG).1Treatment methods include oral pain medications, physical therapy, epidural steroid injection (ESI) and surgery, among others. Both ESI and surgery appear to result in short-term pain relief relative to more conservative measures, yet neither is clearly superior to observation at 1-year follow-up (2,3).

Lumbar epidural steroid injection (LESI) was first suggested as a conservative treatment for radicular pain in 1952 by Robecchi and Capra,4 and it has since become one of the most commonly utilized conservative interventions for radiculopathy.5 Steroids are used to reduce inflammation in the epidural space.6-10 LESI is performed via a transforaminal (TF), caudal (C), or interlaminar (IL) approach in the lumbar spine; these approaches offer different advantages and disadvantages, which may result in different outcomes.11-14 The TF approach is perhaps the most favored because the injection site is adjacent to the nerve root, and only a small volume of medication is required for injection.15 The C route is both the easiest and the safest route and also seems to provide the most favorable analgesic effects. However, this approach requires relatively large volumes of medication and is less specific to the site of pathology.16 Previous studies have described the effectiveness of these methods in the management of radiculopathy.17-22 Magnesium sulfate has not been familiar to anesthesiologists until recently. It has drawn much attention in the field of anesthesiology,23,24 resulting in numerous publications of clinical studies, 25 review articles, and meta-analyses. 26 Based on its diverse roles in cellular functions, magnesium sulfate has been suggested to prevent excitotoxicity by its neuroprotective effects.27 Magnesium can antagonize NMDA receptor channels by blocking calcium influx in a voltage-gated manner. Intravenous administration of magnesium is efficacious in the management of various conditions associated with neuropathic pain. 28,29 Collins and colleagues reported that 70 mg/kg magnesium sulphate infusions in 4 hours for 5 days reduced pain in patients with complex regional pain syndrome. 30 Neuraxial administration of magnesium is an "off-label" use However, animal studies 31,32 showed that intrathecally administered magnesium was free of neurotoxicity, and recent studies have demonstrated the safety of magnesium administration via the epidural route in humans33,34.35 Recently, ozone therapy has emerged as an alternative or additional treatment option for patients with lumbar disc prolapse. Ozone (O 3 ) is an allotropic form of oxygen, primarily known for its ecological properties, industrial application and therapeutic effects. Questions persist concerning its potential toxicity as an oxidant agent versus its reported clinical efficacy. Several mechanisms of action have been proposed to explain the efficacy of ozone therapy including analgesic, anti-inflammatory and oxidant action. The O2-O3 gas mixture injected proximal to the root ganglion is thought to normalize the levels of cytokines and prostaglandins, increase superoxide dismutase levels minimize reactive oxidant species and improve local periganglionic circulation with eutropic effect on the nerve root36,37 Much concern was directed towardsthe contribution of oxidative stress to the pathophysiology of disc prolapse. More and more researchers devote themselves to elucidating the association between oxidative stress and disc degeneration. Antioxidative therapy is suggested as a promising therapeutic approach for preventing or retarding the establishment and progression of disc degeneration. The effect of interventional pain procedures for lumbar disc prolapse on oxidative stress biomarkers such as Glutathione and superoxide dismutase (SOD) remains unknown. 38

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed as having symptomatic lumbar disc prolapse based on the following:

1. Clinical evidence of disc pulge in the form of disc related radicular pain of >3 months duration, not responding to conservative treatment and interfering with daily activities
2. Radiological demonstration of posterolateral lumbar disc pulge by MRI lumbosacral
3. Age range is between 30-80 years

Exclusion Criteria:

The following patients will be excluded from the study:

1. Patients with spinal deformities
2. Patients with a previous history of spinal trauma
3. Patients with previous spinal surgery
4. Patients with radiological evidence of any inflammatory or neoplastic lesion affecting the spinal cord or vertebral column
5. Patients with severe lumbar disc herniation causing lower limb weakness or sphincteric troubles
6. Patient with pain rather than radicular neuropathic pain as Facet osteoarthritis, Sacroiliitis, Hip osteoarthritis, Discogenic, Pyriformis syndrome.
7. Patients with contraindications to interventions (coagulopathy, sepsis, or allergy to the used drugs)
8. Patients with contraindications for MRI examination (e.g., metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body).
9. Pregnant
10. History of G6PD deficiency in patients who are candidates to receive ozone therapy.
11. Suspected spondylodiscitis.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-05 (Estimated); Primary Completion 2021-01-05 (Estimated); Study Completion 2021-04-05 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress biomarkers | 2 weeks post intervention
  (Glutathione (GSH) and superoxide dismutase (SOD))
Pain relief | 3 months post intervention
  Numeric Rating Scale
Disability improvement | 3 months post intervention
  Numeric Rating Scale

SECONDARY OUTCOMES:
Patient satisfaction | 3 months post intervention
  The Short Assessment of Patient Satisfaction (SAPS)

CONTACTS AND LOCATIONS:
Locations (1):
- Wael Fathy Hassan, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided